CLINICAL TRIAL: NCT01919307
Title: Auricular Acupuncture For The Treatment Of Non-Epileptic Seizures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Edward Maa, Chief of the Comprehensive Epilepsy Program, Denver Health and Hospital Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0313
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Convulsion, Non-Epileptic
Keywords: Seizures; Convulsions; Anticonvulsants; Epilepsy; Neurologic
MeSH Terms: conditions — Seizures; Epilepsy; Neurologic Manifestations | interventions — Acupuncture, Ear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Auricular acupuncture (Experimental): Subjects will then receive auricular acupuncture (NADA Protocol) twice weekly for eight consecutive weeks. Subjects will be evaluated for seizure frequency changes by self-reported diary; adverse events; study feasibility; and mental and physiological symptoms at baseline, 12 weeks (completion of acupuncture), and 16 weeks (1 month after treatment follow up, end of study). A single sham procedure will be tested following treatment completion for use in future studies.
  Interventions: Other: Auricular acupuncture

INTERVENTIONS:
Other: Auricular acupuncture — The NADA Protocol for auricular acupuncture will be performed by the PI, a certified NADA protocol practitioner, using sterile, single-use, Seiren 0.22mm, one cm disposable detox needles. Both ears will be sterilized with alcohol swabs. There will be no electrical or other stimulation performed. Needles will be placed subcutaneously with one half twirl upon insertion to the following 5 points (in order per ear): Sympathetic, Shen Men, Kidney, Liver, Lung. Needles will remain in place for 40 minutes and will then be removed in the same order as they were inserted. Needles that become dislodged will be replaced per typical NADA protocol.

SUMMARY:
This feasibility study will determine the tolerability of auricular acupuncture, compliance with self-reported seizure tracking, and the quality of a proposed sham acupuncture protocol to inform the design of a large, multi-center, placebo-controlled, double-blind study to demonstrate the therapeutic effect of auricular acupuncture for the treatment of Non-Epileptic Seizures.

DETAILED DESCRIPTION:
Formerly referred to as "psychogenic" or "pseudo" seizures, Non-Epileptic Seizures (NES) are a physical manifestation of a psychological disturbance and are a type of Somatoform Disorder called a conversion disorder. NES are a significant neurological condition occurring with a prevalence of 2 to 33 per 100,000, similar to that of Multiple Sclerosis. Patients suffering from this phenomenon exhibit seizure-like behavior without electrophysiological correlate, and as would be expected, anti-epileptic drugs (AED) are not effective in treating this disorder. These patients are large consumers of health care resources, are frequently unemployed, require public assistance safety-net programs, and are difficult to properly diagnose without the aid of Epilepsy Monitoring Units (EMU). Furthermore, even after proper diagnosis in an EMU, there is no consensus standard of care therapy for this form of conversion disorder. Most frequently patients are referred for mental health therapy (Cognitive Behavioral Therapy) which is frequently not pursued by the patient due to poor access, poor insight, or stigma.

In a survey of our refractory epilepsy clinic, 68% of respondents are using some form of CAM or Complementary and Alternative Medicine, compared with 39% in a Midwestern population. CAM may offer a solution to access and interest-in-therapy in a population of patients experiencing a high frequency of debilitating events, including NES.

As a complementary and alternative medicine, acupuncture is felt to be a safe and cost-effective therapeutic approach to the treatment of many diseases and symptoms. While the effect of acupuncture for the treatment of epilepsy has been equivocal, studies in the setting of mental health disorders such as post-traumatic stress disorder and anxiety have been promising. Auricular acupuncture has been specifically studied in cocaine dependence, smoking cessation, dental anxiety, and PTSD.

Our interest in acupuncture and NES results from studies that show evidence that acupuncture may improve other conversion disorders presenting as psychogenic movement disorders, or psychogenic erectile dysfunction (16). There also appears to be measurable changes in parasympathetic and sympathetic balance attributable to acupoint stimulation, that may explain anecdotal reports of stress and seizure reduction from acupuncture. It should also be noted that the Vagus Nerve Stimulator, an implantable device that controls medically refractory epileptic seizures, and presumably modulates parasympathetic tone, was first approved as adjunctive therapy in pharmacologically resistant epilepsy by the FDA in 1997 and was later approved for treatment-resistent depression in 2005.

Based on this literature we are conducting an un-blinded treatment trial to establish if auricular acupuncture can effect seizure frequency in NES, and to help design a large double-blind, placebo-controlled clinical trial to determine the efficacy of auricular acupuncture as a treatment for NES. In addition to potentially uncovering an effective treatment for NES, this research will add to our empiric knowledge of acupuncture in conversion disorders such as NES and stimulate further research in acupuncture and NES, both understudied areas.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of non-epileptic seizures, confirmed by ictal routine EEG or ictal video EEG
2. Age 18-75
3. Ability to provide informed consent and comply with study activities
4. > 2 NES per month

Exclusion Criteria:

1. Serious mental health disorder or medical or neurological illness (requiring systemic treatment and/or hospitalization) until subject either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 30 days prior to study entry.
2. Pregnancy, self-discovered pregnancy, lactation, or plans to become pregnant.
3. Inability to distinguish between NES and comorbid epileptic seizures.
4. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
5. Inability or unwillingness of subject or legal guardian/representative to give written informed con-sent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Maa, MD, Principal Investigator — Denver Health
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Auricular Acupuncture
Started | 29
Completed | 20
Not Completed | 9
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Arm/Group | Auricular Acupuncture
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 25
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Completion Rate of Auricular Acupuncture in Patients With NES
Description: Of subjects who receive the first Auricular Acupuncture treatment, we will measure the percentage that goes on to complete the entire 8 week active treatment period.
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Auricular Acupuncture
Number analyzed (Participants) | 29
Participants | 15

2. Secondary Outcome: Adverse Events
Description: We will report the types and rates of any adverse events collected from subject diaries.
Time Frame: 16 Weeks
Measure: Count of Units; unit: Adverse Events
Units Other Than Participants: Adverse Events
Arm/Group | Auricular Acupuncture
Number analyzed (Participants) | 29
Number analyzed (Adverse Events) | 64
Adverse Events
  Nausea | 5
  Dizziness | 4
  Headache | 6
  Pain/Tenderness | 9
  Skin Irritation | 1
  Weakness | 1
  Sleepiness | 3
  Panic/Anxiety | 2
  Seizure | 12
  Hospital Visit | 3
  Withdrawal from Study | 9
  Other | 9

3. Secondary Outcome: Compliance Rates of NES Seizure Diary
Description: For each subject enrolled, we will measure the percentage of diary entries each patient completed over the four month study period.
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: percentage of completed diary entries
Arm/Group | Auricular Acupuncture
Number analyzed (Participants) | 29
percentage of completed diary entries | 90 (8)

4. Secondary Outcome: Trend for Auricular Acupuncture to Reduce NES Frequency
Description: Of subjects completing the 8 week active treatment period, we will compare each subject's 1 month baseline frequency with frequency immediately upon completion of the active treatment period, and at 1 month follow up (3 months after baseline)
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Number of Seizures per Week
Arm/Group | Auricular Acupuncture
Number analyzed (Participants) | 20
Number of Seizures per Week
  Baseline | 15 (16)
  Treatment | 13 (16)
  Washout | 16 (36)

ADVERSE EVENTS:
Time Frame: adverse event data was collected over the course of patient participation, typically 90 days
Arm/Group | Auricular Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes